CLINICAL TRIAL: NCT00830037
Title: Pathobiology of Kidney Disease: Role of Iron
Brief Title: A Clinical Trial of Oral Versus IV Iron in Patients With Chronic Kidney Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by the DSMB based on low chance of finding differences in mGFR slopes, but higher risk of serious adverse events in the IV iron group (aIRR = 1.60)
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK71633; U01DK071633 (NIH); 5U01DK071633-02 (NIH)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Kidney Disease; Iron-deficiency Anemia
Keywords: anemia; iron; kidney disease; progression; glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency; Anemia; Kidney Diseases; Disease Progression | interventions — ferryl iron; Ferric Oxide, Saccharated; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Iron (Experimental)
  Interventions: Drug: IV Iron
- Oral Iron (Active Comparator)
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: IV Iron — IV iron sucrose 200 mg over 2 hours baseline visit, week 2, week 4, week 6 and week 8 for a total of 1000mg total dose. Further cycles of iv iron may be used based on periodic monitoring of iron stores.
  Other Names: Venofer
  Arms: IV Iron
Drug: Ferrous Sulfate — Oral ferrous sulfate 325mg three times daily over 8 weeks. Further cycles of oral iron may be used based on periodic monitoring of iron stores.
  Arms: Oral Iron

SUMMARY:
The long-term goal is to assess the fall in kidney function measured by glomerular filtration rate (GFR) when patients with chronic kidney disease (CKD) are exposed to intravenous iron (IVIR). We hypothesize that in subjects with mild to moderate CKD, infusion of intravenous iron (IVIR), will generate oxidative stress and cause an inflammatory response that will be associated with a more rapid decline in glomerular filtration rate (GFR) compared to oral iron.

DETAILED DESCRIPTION:
Intravenous iron is commonly utilized and is likely a mechanism of renal injury in patients with CKD. This proposal will provide translational data on the role of intravenous iron to progression of kidney disease in patients with CKD. Comparison of IV iron with oral iron will allow testing the hypothesis that IVIR will generate an inflammatory response and albuminuria in the short-term, that will directly lead to a greater rate of fall in GFR, in the long-term, compared to oral iron. We hypothesize that after administration of one gram of IV iron over a course of 8 weeks, renal injury as documented by albuminuria (and fall in GFR) will be increased with IV iron sucrose therapy compared to those randomized to oral iron therapy. A randomized, parallel group, controlled trial will be performed. GFR will be measures every 6 months for two years in 200 participants by iothalamate clearances.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Calculated GFR by MDRD formula < or = 60ml/min/1.73m2. We will use the MDRD formula that incorporates serum creatinine, age, race and sex, but not albumin, and blood urea nitrogen.
* Presence of anemia and iron deficiency. Anemia will be defined as blood hemoglobin concentration <12g/dL and iron deficiency will be defined using National Kidney Foundation/Kidney Disease Outcome Quality Initiative (NFK-K/DOQI) Guidelines as serum ferritin concentration of <100ng/mL or serum transferrin saturation of <25%.

Exclusion Criteria:

* Pregnant or breastfeeding women or women who are planning to become pregnant or those not using a reliable form of contraception (oral contraceptives, condoms, and diaphragms will be considered reliable).
* Known hypersensitivity to iron sucrose (Venofer), iothalamate meglumine (Conray 60, Mallinckrodt) or iodine.
* Anemia that requires RBD transfusion (Hgb <8g/dL) or may potentially need transfusion (active gastrointestinal bleeding). It would be unsafe to withdraw 150 mL blood over the study in such anemic patients.
* Presence of acute renal failure defined as an increase in the baseline serum creatinine concentration of 0.5 mg/dl over 48 hours. This would produce oxidative stress by itself, may give unreliable rate of decline in renal function and may confound results.
* History of IVIR use within 1 month of the study (may confound results of the study if the baseline oxidative stress is increased).
* Evidence of iron overload (serum ferritin >800ng/nl or transferrin saturation >50%)
* Anemia not caused by iron deficiency eg. sickle cell anemia.
* Surgery or systemic or urinary tract infection within 1 month.
* Organ transplant recipient or therapy with immunosuppressive agents. Nasal or inhaled corticosteroids will be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-08; Primary Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD FASN FAHA, Principal Investigator — Indiana University
Locations (1):
- VA Medical Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Iron | Oral Iron
Started | 67 | 69
Completed | 49 | 50
Not Completed | 18 | 19
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Active when terminated by DSMB | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Iron | Oral Iron | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.7) | 67.8 (11.5) | 65.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 50 | 54 | 104
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 27 | 18 | 45
  Hispanic | 2 | 0 | 2
  White | 38 | 51 | 89
eGFR [Mean (Standard Deviation); unit: ml/min per 1.73m2] — Estimated GFR by the four-component MDRD (Modification of Diet in Renal Disease) formula
  ml/min per 1.73m2 | 34.3 (10.2) | 34.7 (10.0) | 34.5 (10.0)
Proteinuria [Number; unit: participants] — Proteinuria was estimated using measurements of urinary protein and creatinine before iron administration at baseline
  participants
    High proteinuria stratum (≥3g/g) | 9 | 9 | 18
    Low proteinuria stratum (<3g/g) | 58 | 60 | 118

OUTCOME MEASURES:

1. Primary Outcome: Mean Rate of Decline in mGFR in the Two Groups - Oral and IV Iron
Description: Plasma clearance of iothalamate was measured by administering an IV bolus of 5 mL of iothalamate meglumine and sampling 2 mL of blood at 0, 5, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, and 300 min after injection. Iothalamate was measured by high-performance liquid chromatography. Plasma clearance was calculated using a two-pool model using validated pharmacokinetic software. The mean modeled iothalamate mGFR slope (e.g., change from baseline to 2 years) in each group (IV iron vs. oral iron) was then calculated after adjustment for baseline log urinary protein/creatinine ratio.
Time Frame: Baseline, 2 years
Population: Modeled iothalamate mGFR slope (e.g., change from baseline to 2 years) was calculated for each group (IV iron vs. oral iron) after adjustment for baseline log urinary protein/creatinine ratio.
Measure: Number; unit: Slope (ml/min per 1.73m2 per year)
Arm/Group | IV Iron | Oral Iron
Number analyzed (Participants) | 67 | 69
Slope (ml/min per 1.73m2 per year) | -4.0 | -3.6
Statistical Analysis 1: Comparison: IV Iron vs Oral Iron; The analysis of the primary outcome was intention to treat, if the patient received at least one dose of the randomized drug (which was the case for each subject). A linear mixed model was used with GFR as the outcome variable. Fixed effects were indicator variables for time (treated as a continuous variable), treatment, and their interaction. Random effects were subject and time with unstructured covariance; statistical inference was made using the maximum likelihood estimator; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis — a = 0.05; Wald test; Mean Difference (Net) = -0.35, 95% CI 2-sided [-2.9 to 2.3]

2. Secondary Outcome: Proteinuria
Description: Proteinuria was estimated using measurements of urinary protein and creatinine before iron administration at baseline and at periodic intervals thereafter. Mean change from baseline log urinary protein/creatinine ratio (g/g) is reported at 2 years.
Time Frame: Baseline, 2 years
Measure: Mean (95% Confidence Interval); unit: g/g
Arm/Group | IV Iron | Oral Iron
Number analyzed (Participants) | 67 | 69
g/g | 0.287 [0.053 to 0.521] | 0.251 [0.019 to 0.484]
Statistical Analysis 1: Comparison: IV Iron vs Oral Iron; The secondary analysis examined the mean change from baseline proteinuria (log protein to creatinine ratio) at 2 years. The between-groups difference in mean change from baseline is reported with a 95% confidence interval and the p-value from the Wald test; Test type: Superiority or Other; p = 0.83, Mixed Models Analysis — a = 0.05; Wald test; Mean Difference (Net) = 0.035, 95% CI 2-sided [-0.294 to 0.365]

ADVERSE EVENTS:
Time Frame: Adverse event data were routinely collected at 2, 4, 6, and 8 weeks after randomization during the treatment phase and again at 3, 6, 12, 18, and 24 months after randomization during the follow-up phase.
Arm/Group | IV Iron | Oral Iron
Serious Adverse Events (participants affected / at risk) | 37/67 | 40/69
Other Adverse Events (participants affected / at risk) | 45/67 | 47/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Iron (N=67) | Oral Iron (N=69)
Skin infection (Infections and infestations) | 7 (11) | 6 (6)
Bone infection (Infections and infestations) | 3 (4) | 2 (7)
Lung infection (Infections and infestations) | 8 (11) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (5)
Sepsis (Infections and infestations) | 5 (5) | 1 (2)
Infections and infestations - other, miscellaneous (Infections and infestations) | 1 (1) | 2 (3)
Heart failure (Cardiac disorders) | 9 (28) | 9 (15)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 8 (9) | 8 (9)
Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 4 (5) | 4 (4)
Pulmonary valve disease (Cardiac disorders) | 2 (3) | 1 (2)
Cardiac disorders - other, miscellaneous (Cardiac disorders) | 5 (6) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 12 (21) | 15 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4) | 5 (6)
Renal and urinary disorders - other, miscellaneous (Renal and urinary disorders) | 3 (3) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, cancer-related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (8) | 4 (4)
Surgical and medical procedures - other, PRBC transfusion (Surgical and medical procedures) | 12 (19) | 12 (17)
Gastrointestinal disorders - other, GI bleed (Gastrointestinal disorders) | 0 (0) | 5 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Retinopathy (Eye disorders) | 1 (5) | 1 (2)
Hypertension (Vascular disorders) | 3 (5) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (3) | 2 (3)
General disorders and administration site conditions - other, miscellanous (General disorders) | 20 (27) | 21 (33)
Renal and urinary disorders - other, end stage renal disease (Renal and urinary disorders) | 6 (6) | 7 (7)
Death NOS (General disorders) | 6 (6) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Iron (N=67) | Oral Iron (N=69)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, new cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chest pain, cardiac (Cardiac disorders) | 0 (0) | 2 (3)
Heart failure (Cardiac disorders) | 3 (4) | 1 (1)
Cardiac disorders - other, miscellaneous (Cardiac disorders) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Metabolism and nutrition disorders - other, new onsent diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - other, miscellaneous (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 9 (10)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders - other, gastroenteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorders - other, miscellaneous (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastrointestinal disorders - other, stool discoloration (Gastrointestinal disorders) | 0 (0) | 10 (10)
Gastrointestinal disorders - other, hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - other, gout (Metabolism and nutrition disorders) | 4 (13) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (5)
Dizziness (Nervous system disorders) | 9 (12) | 9 (10)
Lung infection (Infections and infestations) | 3 (4) | 3 (3)
Infections and infestations - other, miscellaneous (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (8) | 10 (10)
Urinary tract infection (Infections and infestations) | 10 (10) | 4 (5)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 4 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Injury, poisoning and procedural complications - other, traumatic injury (Injury, poisoning and procedural complications) | 2 (2) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Surgical and medical procedures - other, outpatient procedure (Surgical and medical procedures) | 7 (7) | 7 (9)
Non-cardiac chest pain (General disorders) | 1 (1) | 5 (6)
Musculoskeletal and connective tissue disorder - other, leg cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 3 (3)
General disorders and administration site conditions - other, miscellaneous (General disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Vascular disorders - other, venous clot (Vascular disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Nervous system disorders - other, entrapment neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Endocrine disorders - other, thyroid orbitopathy (Endocrine disorders) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - other, rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, thyroid cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
General disorders and administration site conditions - other, drug reaction (General disorders) | 2 (2) | 2 (2)
Injury, poisoning and procedural complications - other, stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - other, access-related (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Skin infection (Infections and infestations) | 3 (4) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No